CLINICAL TRIAL: NCT01575444
Title: Minnesota Community Networks Center for Eliminating Cancer Disparities: Cervical Cancer Screening Project Part C Quantitative
Brief Title: Cervical Cancer Screening Project Part C
Status: Terminated | Type: Observational
Why Stopped: Investigator left University No results are possible
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2010NTLS097
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Cervical Cancer
Keywords: Pap test; HPV testing; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Home based or clinic based HPV test (Pap) collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Home Based Vaginal Collection: Somali women who are randomized for Home based Vaginal Collection will be given a kit to perform the vaginal sample collection for HPV analysis, with detailed written instructions.
- Clinic Based Pap Test Collection: 30 Somali women who are randomized for Standard Clinic Pap Group will be given a list of clinics that they can attend for cervical cancer screening using pap test. Follow-up will be done on test completion with the clinic at 3 months after enrollment.

SUMMARY:
This proposal has been developed through collaboration between the University of Minnesota and New American Community Services (NACS), and the research design is based on a needs assessment conducted by the community partner. The investigators will test the hypotheses that women who are offered home vaginal bio-specimen collection will have higher rate of cervical cancer screening completion than that of women referred for clinic-based Pap test. All participants will be given identical education materials on cervical cancer screening and HPV, currently in use by the Minnesota Sage Program.

DETAILED DESCRIPTION:
The trial will pilot text a protocol for home vaginal bio-specimen collection for human papillomavirus (HPV) testing for cervical cancer screening. The main objective is to estimate the successful screening completion rate among a sample of Somali women who have not undergone cervical cancer screening for three or more years. Women will be randomized to either home vaginal bio-specimen collection or referral to undergo a clinic-based Pap test.

ELIGIBILITY:
Inclusion Criteria:

* Somali female age 25-70 years

  * have lived in the U.S. 10 years or less
  * have not had a Pap test (by self report) in the last 3 years

Exclusion Criteria:

* Women with a self reported past history of any of the following will not be eligible:

  * total hysterectomy
  * cervical cancer
  * active history of cervical dysplasia

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Somali female - Participants may speak Somali or English as their primary language.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of home vaginal bio-specimen collections compared to standard clinic-based Pap test | Within 3 months after Enrollment
  The main outcome will be successful completion of cervical cancer screening by 3 months after enrollment. For the Home Vaginal Biospecimen Collection Group, completion is defined as return of the HPV DNA self-sampling kit by the patient, with a sample suitable for laboratory analysis. In the Clinic Pap Test Group, completion is defined by documentation of Pap test result.

CONTACTS AND LOCATIONS:
Overall Officials: Rahel Ghebre, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States